CLINICAL TRIAL: NCT06477068
Title: Effect of a Medication Reminder Mobile Application on Patients Undergoing Ovarian Stimulation: a Randomized Controlled Trial
Brief Title: Effect of a Medication Reminder Mobile Application
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hung Vuong Hospital (Other)
Responsible Party: Principal Investigator, Thi Thanh Thuy Tran, MD, Hung Vuong Hospital, Hung Vuong Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CS/HV/23/29
Record Dates: First submitted 2024-05-25; First posted 2024-06-27 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Experimental group: Patients undergoing ovarian stimulation in the Infertility Department at Hung Vuong Hospital are prescribed and instructed to inject medication according to the current procedure of the department, in addition to being supported through the "telemedicine medication reminder app on smartphones".
  Control group: Patients undergoing ovarian stimulation in the Infertility Department at Hung Vuong Hospital are prescribed and instructed to inject medication according to the current procedure of the department.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVF Patients (Experimental): Patients undergoes ovarian stimulation for IVF treatment at Hung Vuong Hospital
  Interventions: Combination Product: Mobile medical reminder application

INTERVENTIONS:
Combination Product: Mobile medical reminder application — Experimental group: Patients undergoing ovarian stimulation in the Infertility Department at Hung Vuong Hospital are prescribed and instructed to inject medication according to the current procedure of the department, in addition to being supported through the "telemedicine medication reminder app on smartphones".
  Control group: Patients undergoing ovarian stimulation in the Infertility Department at Hung Vuong Hospital are prescribed and instructed to inject medication according to the current procedure of the department.

SUMMARY:
The goal of this clinical trial is to evaluate of effectiveness when using the "telemedicine medication reminder app on smartphones" at the Infertility Department of Hung Vuong Hospital. The main questions it aims to answer are:

Comparison of the medication forgetting rate between the group of patients using the product and the group of patients not using the app.

Assessment of the level of patient satisfaction when using the app. Comparison of the quantity and quality outcomes of eggs between the group of patients using the app and the group of patients not using the app.

Participants will:

Using or not using " "telemedicine medication reminder app on smartphones" Record the number of cycle cancellations, number of missed doses, satisfaction rates, number of retrieved oocytes, number of mature oocytes, number of immature oocytes, and number of abnormal oocytes.

DETAILED DESCRIPTION:
Goal of SMART:

S Specific: fertility specialists at the Infertility Department of Hung Vuong Hospital, researchers at the Department of Biomedical Engineering - International University - National University of Ho Chi Minh City, and patients at the Infertility Department of Hung Vuong Hospital. Fertility specialists will be responsible for advising and assisting the research team in developing the "telemedicine medication reminder app on smartphones" tailored to the needs and user-friendly for patients. They will support data collection to compare the effectiveness of product usage. Researchers will be responsible for developing and improving the "telemedicine medication reminder app on smartphones" according to the requirements of fertility specialists and patients, as well as analyzing data to evaluate the product's effectiveness.

M Measurable: The effectiveness of the "telemedicine medication reminder app on smartphones" will be compared between the group of patients using the product and the group of patients not using it: Comparison of the medication forgetting rate between the group of patients using the product and the group of patients not using the product.

Evaluation of patient satisfaction level when using the product. Comparison of the quantity and quality outcomes of eggs between the group of patients using the product and the group of patients not using the product.

A Attainable: The Department of Biomedical Engineering has developed numerous telemedicine healthcare products and achieved notable successes, exemplified by the telemedicine blood pressure monitor.

The Infertility Department has a policy to foster scientific research collaboration, aiming to enhance treatment effectiveness and patient satisfaction.

The Infertility Department is a prominent and reputable reproductive support center with a large number of patients, facilitating data collection needs.

R Realistic: The demand for remote monitoring and home healthcare is a legitimate need for patients, especially following the COVID-19 pandemic.

T Time-bound: This research will be conducted over a period of 18 months with specific tasks including 10 months for mobile application development, 6 months for patients recruitment and 2 months for data analysis and interpretation.

ELIGIBILITY:
Inclusion Criteria:

* To eliminate factors that may affect egg quality, we selected patients with good prognosis for the study (18-< 40 years old, undergoing IVF treatment for the first time).
* Indicated for ovarian stimulation for IVF treatment.
* Be able to use a smartphone.
* No underlying diseases: Diabetes mellitus, Increased prolactin, Thyroid dysfunction, and Adrenal disorders.
* Voluntary participate in the study and agree to sign the consent form.

Exclusion Criteria:

* BMI > 30.
* IVF patient with oocyte donation.
* Reduced ovarian reserve.
* Contraindications for using ovarian stimulation drugs.
* Endocrine or metabolic disorders, any underlying diseases (kidney, liver, or heart disease).
* Subjects unwilling to participate in the study.
* Patients who are unable to comply with the study protocol: not using a smartphone, missing appointments for follow-up visits, unable to read or write in Vietnamese.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 387 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Medication non-adherence rate | 6 months
  Comparison of the medication non-adherence rate (in percentage) between the group of IVF patients using the mobile medical reminder application and the group of IVF patients not using the mobile medical reminder application.
  The medication non-adherence rate is calculated as the number of times the medication was forgotten divided by the total number of prescribed medication doses.
  Unit of measure: Percentage (%)
Grading on Mobile Application Rating Scale | 6 months
  Assessment of the mobile medical reminder application quality will be graded following the Mobile Application Rating Scale (MARS). MARS includes a set of questions that are graded by users. Users will rate the app on a scale from 1 to 5. The average MARS score will be used.
  Unit of measure: Quality score (MARS)

SECONDARY OUTCOMES:
Total retrieved oocytes | 6 months
  The number of oocytes retrieved will be recorded and compared between the group of IVF patients using the mobile medical reminder application and the group of IVF patients not using the mobile medical reminder application.
  Unit of measure: Count (number)
Total mature oocytes | 6 month
  The number of retrieved mature oocytes will be recorded and compared between the group of IVF patients using the mobile medical reminder application and the group of IVF patients not using the mobile medical reminder application Unit of measure: Count (number)
Total abnormal oocytes | 6 month
  The number of retrieved abnormal oocytes will be recorded and compared between the group of IVF patients using the mobile medical reminder application and the group of IVF patients not using the mobile medical reminder application Unit of measure: Count (number)

CONTACTS AND LOCATIONS:
Overall Officials: Le-Giang Tran, Ph.D., Principal Investigator — International University, Vietnam National University - Hochiminh City
Locations (1):
- Hung Vuong, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
The research group does not have the ownership of the patient data.